CLINICAL TRIAL: NCT02966652
Title: A Phase 1, Randomised, Open-label, 2-cohort, Cross-over Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of a Native Oral Testosterone Formulation (DITEST) in the Fed and Fasted State and Compared to Testosterone Undecanoate in Adult Men With Primary or Secondary Hypogonadism
Brief Title: Study to Compare DITEST to Testosterone Undecanoate in Adult Men With Hypogonadism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine UK Limited (Industry)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other); Simbec Research (Industry); Voet Consulting (Industry); EMAS Pharma (Industry); Medical Matters International Ltd (Industry); Brush Clinical Research Ltd. (Industry); Manchester University NHS Foundation Trust (Other Government); Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DITEST-001
Record Dates: First submitted 2016-09-26; First posted 2016-11-17 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-10

CONDITIONS: Male Hypogonadism
Keywords: Male; Hypogonadism; Primary; Secondary; Androgen deficiency
MeSH Terms: conditions — Eunuchism; Hypogonadism; Neoplasm Metastasis | interventions — testosterone undecanoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testosterone undecanoate (Active Comparator): Cohort 1: single dose of 120 mg (3 x 40 mg) DITEST followed by a single dose of 80 mg (2 x 40 mg) testosterone undecanoate or a single dose of 80 mg (2 x 40 mg) testosterone undecanoate followed by single dose of 120 mg (3 x 40 mg) DITEST. The two treatments are separated by a minimum of a 7-day washout period, with both treatments given in the fed state.
  Interventions: Drug: DITEST; Drug: Testosterone undecanoate
- DITEST (Experimental): Cohort 2: single dose of 200 mg (5 x 40 mg) DITEST (fed) followed by a single dose of 200 mg DITEST (fasted) or a single dose of 200 mg DITEST (fasted) followed by single dose of 200 mg (5 x 40 mg) DITEST (fed). The two treatments are separated by a minimum of a 7-day washout period.
  Interventions: Drug: DITEST

INTERVENTIONS:
Drug: DITEST — Lipid formulation of native oral testosterone.
Drug: Testosterone undecanoate — Generic treatment for patients with primary or secondary male hypogonadism
  Arms: Testosterone undecanoate

SUMMARY:
DITEST is an oral formulation of native testosterone for the treatment of androgen deficiency in men. The study was a Phase 1 clinical study in hypogonadal men, defined according to FDA and Endocrine Society Guidelines, designed to evaluate the pharmacokinetic (PK) characteristics of DITEST, and to assess the safety and tolerability of DITEST in the target population.

DETAILED DESCRIPTION:
There is an unmet need for a native oral testosterone therapy for men with androgen (testosterone) deficiency. Ideally such a treatment should have reproducible PK, does not need to be taken with fatty meals, can be taken once or twice daily, and provides physiological exposure to testosterone. This Phase 1, randomised, open-label, 2-cohort, cross-over study was therefore designed to evaluate the PK characteristics of DITEST in both the fed and fasted states according to FDA guidelines, and to assess the safety and tolerability of DITEST in the target population.

The study was conducted in male subjects from 18 to 80 years of age requiring testosterone replacement therapy for primary or secondary hypogonadism. The study was a randomised, active control, single dose, 2-way cross-over study in 2 cohorts. In each cohort subjects who meet the entry criteria at screening and baseline were randomised to one of 2 sequences:

Cohort 1: single dose of 120 mg (3 x 40 mg) DITEST followed by a single dose of 80 mg (2 x 40 mg) testosterone undecanoate (TU) or a single dose of 80 mg TU followed by single dose of 120 mg DITEST. The two treatments were separated by a minimum of a 7-day washout period, with both treatments given in the fed state.

Cohort 2: single dose of 200 mg (5 x 40 mg) DITEST (fed) followed by a single dose of 200 mg DITEST (fasted) or a single dose of 200 mg DITEST (fasted) followed by single dose of 200 mg DITEST (fed). The two treatments were separated by a minimum of a 7-day washout period.

13 subjects were recruited into cohort 1 and 12 subjects were recruited into cohort 2, resulting in a total of 25 subjects being administered study medication in this study. Subjects were not recruited into Cohort 2 until the results of subjects treated in Cohort 1 had been evaluated (this review was to determine if the intended dose for Cohort 2 needed to be adjusted). No other testosterone treatments were allowed for the duration of the study (including the washout periods).

Each subject was required to attend the study centre for a minimum of either 4 or 5 visits: a screening assessment, an evaluation of baseline testosterone levels after the washout period from the subject's current medication (only for subjects currently on testosterone replacement therapy), both dosing days, and a follow-up visit at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged 18 to 80 years.
* Diagnosis of primary testicular failure or secondary hypogonadism due to known pituitary disease or congenital deficit.
* Body mass index (BMI) >18kg/m2 and <35kg/m2
* Testosterone level <8nmol/L after washout of current testosterone treatment, if applicable.
* Normal prostate specific antigen (PSA) levels based on the age of the subject.
* Provision of written informed consent and able to participate in the study and abide by the study restrictions.

Exclusion Criteria:

* Subjects with a past history of, or current prostate cancer, male breast cancer or hepatic neoplasm.
* Subjects with a history of or current myocardial infarction (MI), unstable cardiovascular disease, or clinically relevant findings on the screening electrocardiogram (ECG) (as determined by the investigator)
* Subjects with a history of or current alcohol abuse (consumption of more than 28 units per weekweek: 1 unit equals 25mL single measure of whisky (ABV 40%), a third of a pint of beer (ABV 5-6%) or half a standard (175 mL) glass of red wine (ABV 12%).
* Subjects with other unstable or inadequately treated endocrine conditions.
* Haematocrit levels >0.5 at baseline
* Subjects with poor dental hygiene that would interfere with the collection of saliva samples or contaminate them with blood.
* Subjects with any severe co-morbidity or with any significant medical or psychiatric conditions that in the opinion of the investigator would preclude participation in the trial.
* Participation in another clinical trial or an investigation or licensed drug or device within the 3 months prior to inclusion in this study.
* Allergic to any of the ingredients in the DITEST capsule, particularly sesame oil, or to any components of testosterone undecanoate capsules, particularly castor oil.
* Subjects with a known intolerance to alcohol (e.g. flushing) or ethnic populations at high risk of alcohol dehydrogenase (ADH) enzyme polymorphism with potential to impair metabolism of benzyl alcohol and ethanol, both of which are contained in the DITEST formulation.
* Meeting any of the contraindications for testosterone undecanoate, as detailed in the Summary of Product Characteristics (SmPC) of the comparator product.
* Subjects who are unable to consume the standard high-fat breakfast.
* Subjects who have donated blood or plasma in the previous 3 months prior to screening.
* Any subjects taking a concomitant medication known to enhance or inhibit the action of p450 CYP3A4 (rifampicin, barbiturates, carbamazepine, dichloralphenazone, phenylbutazone, phenytoin or primidone).

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

PRIMARY OUTCOMES:
Testosterone serum concentrations - Peak Plasma Concentration (Cmax) | Study day 0 to Study Day >7 (sampling time points at -0.5, 0.25 [120mg and TU arms only], 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8 and 10 hours post-Investigational Medicinal Product (IMP) administration, on each visit date)
  Testosterone serum concentrations after administration of a single dose of 120mg or 200mg DITEST and 80mg testosterone undecanoate in the fed state, as measured by the primary PK parameter of Cmax.
Testosterone serum concentrations - Area under the serum testosterone concentration-time curve from time 0-10 (AUC(0-10)) | Study day 0 to Study Day >7 (sampling time points at -0.5, 0.25 [120mg and TU arms only], 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8 and 10 hours post-IMP administration, on each visit date)
  Testosterone serum concentrations after administration of a single dose of 120mg or 200mg DITEST and 80mg testosterone undecanoate in the fed state, as measured by the primary PK parameter of AUC.

SECONDARY OUTCOMES:
Testosterone serum concentrations - Peak serum testosterone Concentration (Cmax) | Study day 0 to Study Day >7 (sampling time points at -0.5, 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8 and 10 hours post-IMP administration, on each visit date)
  Testosterone serum concentrations after 200mg dose of DITEST in the fed and fasted states, as measured by the primary PK parameter of Cmax.
Testosterone serum concentrations after 200mg dose - Area under the serum testosterone concentration-time curve (AUC 0-10) | Study day 0 to Study Day >7 (sampling time points at -0.5, 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8 and 10 hours post-IMP administration, on each visit date)
  Testosterone serum concentrations after 200mg dose of DITEST in the fed and fasted states, as measured by the primary PK parameter of AUC (0-10)
Adverse events | Through study completion - a maximum of 84 days.
  Adverse events (AEs) observed throughout the study.
Vital signs | Through study completion - a maximum of 84 days.
  Observed changes in vital signs data during the course of the study.
Electrocardiogram (ECG) | Through study completion - a maximum of 84 days.
  Observed changes in ECG data during the course of the study.
Safety Laboratory Data | Through study completion - a maximum of 84 days.
  Observed changes in Safety Laboratory data during the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: J Newell-Price, MA, PhD, Principal Investigator — University of Sheffield
Locations (1):
- Sheffield Teaching Hospital - Royal Hallamshire Hospital, Sheffield, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No